CLINICAL TRIAL: NCT00707304
Title: FORTIS-M: A Phase 3, Randomized, Double-blind, Placebo-controlled Study of Oral Talactoferrin in Addition to Best Supportive Care in Patients With Non-small Cell Lung Cancer Who Have Failed Two or More Prior Treatment Regimens
Brief Title: Safety and Efficacy of Talactoferrin in Previously Treated Patients With Non-small Cell Lung Cancer
Acronym: FORTIS-M
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LF-0207; NCT00937209 (obsolete NCT alias)
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Talactoferrin; Dendritic Cell Recruiter and Activator; Immunomodulatory agent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — talactoferrin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Talactoferrin alfa (talactoferrin or TLF, also known as recombinant human lactoferrin, rhLF or talactoferrinum alfa) is a recombinant version of the glycoprotein expressed in and purified from Aspergillus niger var. awamori. Talactoferrin is structurally and functionally similar to native human lactoferrin. The structural equivalence of talactoferrin to native human lactoferrin has been demonstrated by a comparison of the 3-dimensional structure, molecular weight, biological activity and other physicochemical properties, and is known to differ only in the nature of glycosylation.
  Interventions: Drug: Talactoferrin
- 2 (Placebo Comparator): Placebo contains the same phosphate-based buffer used as the diluent for the talactoferrin solution. In addition, the placebo will contain FD&C/EU grade dyes suitable for oral use to mimic the color of the vialed drug product.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Talactoferrin — Oral, 1.5 grams twice per day
  Other Names: talactoferrin alfa; TLF; recombinant human lactoferrin; rhLF
  Arms: 1
Drug: Placebo — Oral, twice per day
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether talactoferrin can improve overall survival in patients with non-small cell lung cancer (NSCLC) who have been previously treated with two or more regimens.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB or IV NSCLC
* Failed at least 2 prior systemic anti-cancer regimens for advanced or metastatic NSCLC
* At least one target lesion that is unirradiated and measurable by RECIST
* Adequate hematologic, renal and hepatic function
* ECOG 0, 1, or 2
* Able to understand and sign an Informed Consent

Exclusion Criteria:

* Presence of brain metastases, unless the patient received brain irradiation, including adequate stereotactic radiosurgery, at least 4 weeks prior to randomization, and is stable, asymptomatic, and off steroids for at least 3 weeks prior to randomization
* Any gastrointestinal tract disease or other medical condition resulting in the inability to take oral medications
* History of other malignancies except: (i) adequately treated basal or squamous cell carcinoma of the skin; (ii) curatively treated, a) in situ carcinoma of the uterine cervix, b) prostate cancer, or c) superficial bladder cancer; or (iii) other curatively treated solid tumor with no evidence of disease for ≥ 5 years
* Uncontrolled ischemic heart disease, or uncontrolled symptomatic congestive heart failure
* Serious active infection
* Psychiatric illness/ social situations that would limit study compliance
* Other uncontrolled serious chronic disease or conditions that in the investigator's opinion could affect compliance or follow-up in the protocol
* Concurrent radiotherapy to any site or radiotherapy within 4 weeks prior to randomization or previous radiotherapy to the target lesion sites (the sites that are to be followed for determination of a response)
* Known HIV positive or on active anti-retroviral therapy
* Known Hepatitis B surface antigen positive or hepatitis C positive
* Receipt of any investigational medication within 4 weeks prior to randomization
* Pregnant or lactating patients, or fertile female patients with a positive pregnancy test, or fertile female patients unwilling to use adequate contraception during treatment and 30 days after completion of treatment
* Sexually active male patients unwilling to practice contraception while participating on the study and up to 30 days after completion of treatment
* Legal incapacity or limited legal capacity, unless authorization is granted by a legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | After the occurence of the required number of events

SECONDARY OUTCOMES:
Progression free survival | At time of final analysis
Objective response and disease stablization rate | At time of final analysis
Safety and tolerability | At time of final analysis

CONTACTS AND LOCATIONS:
Locations (189):
- United States (29):
  - Desert Oasis Cancer Center, Casa Grande, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - University of Colorado Hospital, Aurora, Colorado
  - Pasco Pinellas Cancer Center, New Port Richey, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Central Indiana Cancer Centers, Greenfield, Indiana
  - Kansas City Cancer Center, LLC, Overland Park, Kansas
  - NCI, CCR, The Waren Grant Magnuson Clinical Center, Bethesda, Maryland
  - Newland Medical Associates, Southfield, Michigan
  - Minnesota Oncology and Hematology, PA, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - NH Oncology-Hematology, PA, Hooksett, New Hampshire
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Alamance Regional Medical Center, Burlington, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Legacy Pharma Research, Bismarck, North Dakota
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Kaiser Group Health, Portland, Oregon
  - Texas Oncology, Dallas, Texas
  - Texas Oncology, Fort Worth, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Oncology & Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Salem, Virginia
  - Cancer Care Northwest, Spokane, Washington
- Australia (5):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Townsville Hospital, Townsville, Queensland
  - The Queen Elisabeth Hospital, Woodville South, South Australia
  - Epworth Healthcare, Richmond, Victoria
- Bulgaria (5):
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven, Pleven
  - DDODIU-Plovdiv, EOOD, Aleksandur Stamboliyski, Plovdiv
  - DDODIU-Plovdiv, EOOD, Plovdiv, Plovdiv
  - DDODIU - Sofia District EOOD, Sofia
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Mount Sinai Hospital, Toronto, Ontario
  - Hôtel-Dieu de Lévis, Lévis, Quebec
  - Gerald Bronfman Centre for Clinical Research in Oncology, Montreal, Quebec
- Czechia (9):
  - Pardubicka krajska nemocnice, a.s., Pardubice, Pardubice
  - Fakultni nemocnice Na Bulovce, Budinova, Prague
  - Oblastni nemocnice Pribram, a.s., Příbram, Pribram
  - Institut Onkologie a Rehabilitace Na Plesi, Nová Ves pod Pleší
  - Vitkovicka nemocnice a.s., Ostrava
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
  - Fakultni nemocnice v Motole, s.p., Prague
  - Nemocnice Tabor, a.s., Tábor
- France (17):
  - CHU Angers, Angers, Angers Cedex
  - Centre Francois Baclesse, Caen, Caen Cedex
  - Centre d'Oncology de Gentilly, Cedex, Cedex
  - Hopital Cardiologique, Chru Lille, Lille, Cedex
  - CHU Pontchaillou, Rennes, Cedex
  - CRLCC René Gauducheau, Saint-Herblain, Cedex
  - CLCC Paul Strauss, Strasbourg, Cedex
  - Hopital Larrey, Toulouse, Cedex
  - Centre Hospitalier du Mans, Le Mans, Le Mans Cedex
  - Centre Léon Berard, Lyon, Lyon
  - Centre Catherine de Sienne, Eric Tabarly, Nantes
  - Hôpital Saint-Antoine, Paris, Paris
  - Hopital Maison Blanche, Reims, Reims
  - CHU de Nancy, Hopital de Brabois, Vandœuvre-lès-Nancy, Vandoeuvre Les Nancy
  - Hopital Morvan, Brest
  - Hopital Sainte Marguerite, Marseille
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (12):
  - Praxis fuer interdisziplinaere Onkologie, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Mannheim, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen - PS, Erlangen, Bavaria
  - Asklepios Fachkliniken Muenchen-Gauting, Gauting, Bavaria
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg, Heidelberg
  - Gemeinschaftspraxis fuer Haematologie Onkologie, Wiesbaden, Hesse
  - Universitaetsklinikum Goettingen, Göttingen, Lower Saxony
  - St. Johannes Hospital - PS, Dortmund, North Rhine-Westphalia
  - Staedt. Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle, Saxony-Anhalt
  - Krankenhaus Grosshansdorf, Woehrendamm, Schleswig-Holstein
  - Zentralklinik Bad Berka, Bad Berka, Thuringia
- Greece (6):
  - General Hospital of Athens "Sotiria", Athens, Athens
  - University Hospital of Heraklio, Crete, Crete
  - General Hospital of Chania 'Ag. Georgios', Mourniés, Crete
  - University Hospital of Larissa, Mezourlo, Larissa
  - University General Hospital of Patras, Rio, Patras
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Hungary (8):
  - Semmelweis Egyetem, Budapest, Budapest
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest, Budapest
  - Miskolc Megyei Jogu Varos Onkormanyzat Miskolci Egeszsegugyi, Csabai Kapu, Miskolc
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc, Miskolc
  - Szabolcs-Szatmar Bereg Megyei Josa Andras Oktato Korhaz, Nyiregyháza, Nyiregyháza
  - Fejer Megyei Szent Gyorgy Korhaz, Seregelyesi, Szekesfehervar
  - Torokbalinti Tudogyogyintezet, Törökbálint, Torokbalint
  - Zala Megyei Korhaz, Zalaegerszeg, Zalaegerszeg
- India (16):
  - King George Hospital, Vishakhapattanam, Andhhra Pradesh
  - Apollo Hospital, Hyderabad, Andhra Pradesh
  - Indo-American Cancer Institute and Research Center, Hyderabad, Andhra Pradesh
  - Kidwai Institute of Oncology, Bangalore, Karnataka
  - M. S. Ramaiah Memorial Hospital, Bangalore, Karnataka
  - A.J. Medical College Hosptial, Mangalore, Karnataka
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - P.D. Hinduja Nat. Hospital & Med. Research Centre, Mumbai, Maharashtra
  - Kaushalya Medical Foundation Trust Hospital, Mumbai, Maharashtra
  - Cancer Care Clinic, Nagpur, Maharashtra
  - Shatabdi Hospital, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Center, Pune, Maharashtra
  - Searoc Cancer Hospital, Jaipur, Rajasthan
  - Mahaveer Cancer Hospital and Research Centre, Jaipur, Rajasthan
  - Dr. Kamakshi Memorial Hospital Pvt Ltd, Chennai, Tamil Nadu
  - Christian Medical College Hospital, Vellore, Tamil Nadu
- Italy (9):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I, Ancona, AN
  - CRO Centro di Riferimento Oncologico di Aviano, Aviano, Aviano
  - Istituto per la Ricerca e la Cura del Cancro, Candiolo, Candiolo/TO
  - Azienda Ospedaliera Istituti Ospitalieri di Cremona, Cremona, Cremona
  - Ospedale Versilia, Lido di Camaiore, LU
  - Istituto Nazionale Tumori, Milan, MI
  - Azienda Ospedaliera San Gerardo, Monza, MI
  - Azienda Ospedaliera San Camillo Forlanini, Roma, RM
  - Ospedale Mater Salutis, Legnago, VR
- Latvia (4):
  - Dr. Anna Levcenko GP and Internist Practice, Daugavpils
  - Piejuras Hospital, Liepāja
  - Riga Eastern Clinical University Hospital, Riga
  - P. Stradina Clinical University Hospital, Riga
- Malaysia (4):
  - Nilai Cancer Institute (NCI Cancer Hospital), Negeri Sembilan, Darul Khusus
  - Lam Wah Ee Hospital, Pulau Pinang, Georgetown,
  - Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
- Philippines (3):
  - St. Luke's Medical Center, Quezon City, Quezon City
  - Manila Doctors Hospital, Manila
  - Lung Center of the Philippines, Quezon City
- Poland (6):
  - Akademickie Centrum Kliniczne - Szpital AM w Gdansku, Gdansk, Gdansk
  - Nzoz Vesalius, Krakow, Krakow
  - Miedziowe Centrum Zdrowia S.A., Lubin, Lubin
  - NZOZ Olsztynski Osr. Onkologiczny "Kopernik" Sp.z o.o, Olsztyn, Olsztyn
  - Specjalistyczny Szpital im. Prof. A. Sokolowskiego, Szczecin, Szczecin
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw, Warszawa
- Romania (6):
  - Spitalul Judetean de Urgenta Braila, Brăila, Brăila County
  - S.C. Ianuli Med Consult S.R.L., Bucharest, București
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj-Napoca, Str. Republicii Nr. 34-36, Cluj-Napoca
  - Spitalul Judetean de Urgenta "Sf. Ioan cel Nou" Suceava, Suceava, Suceava
  - Spitalul Judetean de Urgenta "Dr. Constantin Opris", Baia Mare
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj-Napoca, Cluj-Napoca
- Russia (7):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk, Arkhangelskaya oblast
  - SHI Altay Regional Oncology Dispensary, Barnaul, Barnaul
  - CCH #2 n.a. N. A. Semashko of LLC "Russian Railways", Moscow, Moscow
  - City Clinical Hospital #1, Novosibirsk, Novosibirsk Oblast
  - Perm Territorial Oncology Dispensary, Perm, Perm Krai
  - SEIHPE "Saint Petersburg SMU RosZdrav n.a. I.I.Pavlov", Saint Petersburg, Sankt-Peterburg
  - Oncology Dispensary #2 of Krasnodar Region, Dagomysskaya Str., Sochi
- Singapore (4):
  - National Cancer Centre, Hospital Drive, Singapore
  - Parkway Cancer Centre, Mount Elizabeth, Singapore
  - Medical Oncology Centre, Napier Road, Singapore
  - John Hopkins Singapore International Medical Centre, Singapore
- South Korea (8):
  - Chonnam National University Hwasun Hospital, Hwasun Up, Chonnam
  - National Cancer Center, Ilsandong-gu, Goyang
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Samsung Medical Center, Gangnam-Gu, Seoul
  - Seoul National University Hospital, Jongno-gu, Seoul
  - Korea University Anam Hospital, Seongbuk-gu, Seoul
  - Asan Medical Center, Songpa-gu, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Paldal-gu, Suwon Gyeonggi-do
- Spain (5):
  - H Mutua de Terrassa, Barcelona, Barcelona
  - HU Virgen de las Nieves, Granada, Granada
  - Fundacion Jimenez Diaz, Madrid, Madrid
  - HGU La Paz, Madrid, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Pamplona
- Taiwan (6):
  - Changhua Christian Hospital, Changhua, Changhua
  - Kaohsiung Veterans General Hospital, Kaohsiung City, Kaohsiung
  - Taichung Veterans General Hospital, Taichung, Taichung
  - National Cheng Kung University Hospital, Tainan, Tainan
  - Taipei Veterans General Hospital, Taipei, Taipei
  - Chang-Gung Memorial Hospital, Linkou Branch, Toayuan, Toayuan
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty, Ankara, Ankara
  - Gaziantep University Medical Faculty, Gaziantep, Gaziantep
  - Istanbul Bilim University Medical Fac., Istanbul
  - Ege University Medical Faculty, Izmir
- United Kingdom (12):
  - Bristol Haematology & Oncology Centre, Bristol, Brist
  - Guy's & St Thomas' NHS Foundation Trust, London, Gt Lon
  - Christie Hospital, Manchester, Gt Man
  - Southampton General Hospital, Southampton, Hants
  - Castle Hill Hospital, Cottingham Hull, Hull
  - University Hospital of South Manchester NHS Foundation Trust Wythenshawe Hospital, Wythenshawe, Manchester
  - Singleton Hospital, Swansea, S Glam,
  - University Hospital of North Staffordshire, Stoke-on-Trent, Staffs
  - Wolverhampton New Cross Hospital, Wolverhampton, Staffs
  - Beatson West of Scotland Cancer Centre, Glasgow, Strath
  - Ninewells Hospital, Dundee, Tays
  - University Hospital of Coventry and Warwickshire, Coventry, Warwks